CLINICAL TRIAL: NCT03636451
Title: Assessing the Effect of Paracervical Block Volume on Pain Control for Dilation and Curettage: a Randomized Controlled Trial
Brief Title: Effect of Paracervical Block Volume on Pain Control for Dilation and Curettage.o
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: Society of Family Planning (Other); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Sheila Mody, Principal Investigator, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 180999.o; NCT03736681 (obsolete NCT alias)
Record Dates: First submitted 2018-08-13; First posted 2018-08-17 (Actual); Results first posted 2023-04-20 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-03

CONDITIONS: Abortion, Spontaneous; Abortion in First Trimester; Pain Uterus; Abortion Early; Abortion, Missed
Keywords: Dilation & curettage; Paracervical block
MeSH Terms: conditions — Abortion, Spontaneous; Abortion, Missed; Dilatation, Pathologic | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This is a double center, randomized, 2 arm (1:1), single blinded clinical trial comparing pain control at the time of cervical dilation with two different paracervical blocks in women undergoing D&C in the first trimester for either surgical abortion or miscarriage management.
Who Masked: Participant, Outcomes Assessor
Masking Description: The study coordinator, who will be blinded to the intervention, will pick the designated sealed, opaque envelope containing the type of paracervical block and hand it to the physician performing the procedure. The physician will then open the envelope and prepare the designated paracervical block, as it is standard practice for physicians to prepare their own paracervical blocks prior to performing any D&C in-clinic. The paracervical block will contain 2U Vasopressin, 2cc of 8.4% sodium bicarbonate, and either 1% lidocaine or 0.5% lidocaine, depending on the study group. The physician will bring the paracervical block into the clinic room where the procedure will be performed on a covered tray. The physician will perform the standardized procedure for the D&C, and the study coordinator will assess pain control during the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 40cc buffered 0.5% lidocaine with 2 units of vasopressin paracervical block (Experimental): 40c buffered 0.5% lidocaine with 2 units of vasopressin paracervical block with dilation and curettage under minimal sedation
  Interventions: Drug: 40cc buffered 0.5% lidocaine with 2 units of vasopressin paracervical block
- 20cc 1% lidocaine with 2 units of vasopressin paracervical block (Active Comparator): 20cc 1% lidocaine with 2 units of vasopressin paracervical block with dilation and curettage under minimal sedation
  Interventions: Drug: 20cc 1% lidocaine with 2 units of vasopressin paracervical block

INTERVENTIONS:
Drug: 40cc buffered 0.5% lidocaine with 2 units of vasopressin paracervical block — Women undergoing D&C in the first trimester for either surgical abortion or miscarriage management will receive 40cc buffered 0.5% lidocaine with 2 units of vasopressin paracervical block before cervical dilation.
  Other Names: 40cc
  Arms: 40cc buffered 0.5% lidocaine with 2 units of vasopressin paracervical block
Drug: 20cc 1% lidocaine with 2 units of vasopressin paracervical block — Women undergoing D&C in the first trimester for either surgical abortion or miscarriage management will be randomly assigned to receive 20cc 1% lidocaine with 2 units of vasopressin paracervical block before cervical dilation.
  Other Names: 20cc
  Arms: 20cc 1% lidocaine with 2 units of vasopressin paracervical block

SUMMARY:
The investigators are conducting a study on pain control for dilation and curettage (D&C). Participants are eligible to enroll if they are a planning to have a D&C in a participating clinic. The investigators are studying how different ratios of medication to liquid affect pain when injected around the cervix. Both potential methods use the same dose of medication, though researchers would like to know which one works better. To be in this study, participants must be over the age of 18 with an early pregnancy loss or undesired pregnancy measuring less than 12 weeks gestation undergoing D&C while awake in clinic.

DETAILED DESCRIPTION:
Dilation and Curettage (D&C) is often performed in the first trimester for surgical abortion and management of miscarriage and can be painful for patients before and after the procedure. Most procedures are performed while the patient is awake or with minimal sedation in the clinic setting, and a key component of pain control is the paracervical block, or injecting lidocaine into the tissue around the cervix. A paracervical block with 20cc of 1% buffered lidocaine has been proven to provide superior pain control than a sham paracervical block. However, many providers often use similar doses of lidocaine in a higher volume to improve pain control. At University of California, San Diego (UCSD) and University of California, Los Angeles (UCLA), some providers routinely use a 20cc of 1% buffered lidocaine block and some routinely use a 40cc of 0.5% buffered lidocaine block. This practice has not been studied in a randomized controlled trial. The purpose of this study is to compare pain control during D&C with a 20cc 1% buffered lidocaine with vasopressin paracervical block compared to a 40cc 0.5% buffered lidocaine with vasopressin paracervical block.

An inclusion criterion for this study is that patients must specifically be referred to family planning clinics at UCSD and UCLA for an in-clinic D&C. Therefore, the D&C is a required procedure for both study groups. The only difference in care between the study groups will be which paracervical block they receive.

ELIGIBILITY:
Inclusion Criteria:

1. Women over the age of 18 presenting to UC San Diego and UC Los Angeles
2. Undesired pregnancy or missed abortion < 11 weeks 6 days gestation
3. Must speak English or Spanish
4. Desire surgical termination of pregnancy or management of miscarriage in clinic

Exclusion Criteria:

1. Women with a diagnosis of inevitable or incomplete abortion
2. Desire for general anesthesia or IV sedation
3. Chronic pain conditions
4. Any medical comorbidities that are a contraindication to performing the procedure in the clinic setting
5. Allergy to or refusal of ketorolac, oral Versed, or a paracervical block
6. If they have taken any pain medications the day of presentation to clinic
7. If they have taken Misoprostol the day of presentation to clinic

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2022-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila K Mody, MD MPH, Principal Investigator — UCSD Department of Ob/Gyn and Reproductive Sciences
Locations (2):
- United States (2):
  - Villa La Jolla Clinic, La Jolla, California
  - UCSD Medical Offices South, San Diego, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman A. Pain control in first trimester surgical abortion. Cochrane Database Syst Rev. 2009 Apr 15;2009(2):CD006712. doi: 10.1002/14651858.CD006712.pub2. PMID 19370649
- [Background] Renner RM, Jensen JT, Nichols MD, Edelman AB. Pain control in first-trimester surgical abortion: a systematic review of randomized controlled trials. Contraception. 2010 May;81(5):372-88. doi: 10.1016/j.contraception.2009.12.008. Epub 2010 Jan 27. PMID 20399943
- [Background] Meckstroth KR, Mishra K. Analgesia/pain management in first trimester surgical abortion. Clin Obstet Gynecol. 2009 Jun;52(2):160-70. doi: 10.1097/GRF.0b013e3181a2b0e8. PMID 19407522
- [Background] Belanger E, Melzack R, Lauzon P. Pain of first-trimester abortion: a study of psychosocial and medical predictors. Pain. 1989 Mar;36(3):339-350. doi: 10.1016/0304-3959(89)90094-8. PMID 2710563
- [Background] Rawling MJ, Wiebe ER. Pain control in abortion clinics. Int J Gynaecol Obstet. 1998 Mar;60(3):293-5. doi: 10.1016/s0020-7292(97)00254-3. No abstract available. PMID 9544719
- [Background] Stubblefield PG. Control of pain for women undergoing abortion. Suppl Int J Gynecol Obstet. 1989;3:131-40. doi: 10.1016/0020-7292(89)90113-6. PMID 2686702
- [Background] Pud D, Amit A. Anxiety as a predictor of pain magnitude following termination of first-trimester pregnancy. Pain Med. 2005 Mar-Apr;6(2):143-8. doi: 10.1111/j.1526-4637.2005.05030.x. PMID 15773879
- [Background] O'Connell K, Jones HE, Simon M, Saporta V, Paul M, Lichtenberg ES; National Abortion Federation Members. First-trimester surgical abortion practices: a survey of National Abortion Federation members. Contraception. 2009 May;79(5):385-92. doi: 10.1016/j.contraception.2008.11.005. Epub 2008 Dec 11. PMID 19341852
- [Background] Grimes DA, Cates W Jr. Deaths from paracervical anesthesia used for first-trimester abortion, 1972-1975. N Engl J Med. 1976 Dec 16;295(25):1397-9. doi: 10.1056/NEJM197612162952503. PMID 980095
- [Background] Renner RM, Nichols MD, Jensen JT, Li H, Edelman AB. Paracervical block for pain control in first-trimester surgical abortion: a randomized controlled trial. Obstet Gynecol. 2012 May;119(5):1030-7. doi: 10.1097/AOG.0b013e318250b13e. PMID 22525915
- [Background] Renner RM, Edelman AB, Nichols MD, Jensen JT, Lim JY, Bednarek PH. Refining paracervical block techniques for pain control in first trimester surgical abortion: a randomized controlled noninferiority trial. Contraception. 2016 Nov;94(5):461-466. doi: 10.1016/j.contraception.2016.05.005. Epub 2016 May 25. PMID 27235677
- [Background] Jensen MP, Chen C, Brugger AM. Interpretation of visual analog scale ratings and change scores: a reanalysis of two clinical trials of postoperative pain. J Pain. 2003 Sep;4(7):407-14. doi: 10.1016/s1526-5900(03)00716-8. PMID 14622683
- [Background] Rowbotham MC. What is a "clinically meaningful" reduction in pain? Pain. 2001 Nov;94(2):131-132. doi: 10.1016/S0304-3959(01)00371-2. No abstract available. PMID 11690725
- [Background] Todd KH, Funk KG, Funk JP, Bonacci R. Clinical significance of reported changes in pain severity. Ann Emerg Med. 1996 Apr;27(4):485-9. doi: 10.1016/s0196-0644(96)70238-x. PMID 8604867
- [Background] Kroenke K, Spitzer RL, Williams JB, Monahan PO, Lowe B. Anxiety disorders in primary care: prevalence, impairment, comorbidity, and detection. Ann Intern Med. 2007 Mar 6;146(5):317-25. doi: 10.7326/0003-4819-146-5-200703060-00004. PMID 17339617
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Derived] Crouthamel B, Economou N, Averbach S, Rible R, Kully G, Meckstroth K, Mody SK. Effect of Paracervical Block Volume on Pain Control for Dilation and Aspiration: A Randomized Controlled Trial. Obstet Gynecol. 2022 Aug 1;140(2):234-242. doi: 10.1097/AOG.0000000000004862. Epub 2022 Jul 6. PMID 35852274
- See also: Guttmacher Institute: Facts on Induced Abortion Worldwide — https://www.guttmacher.org/fact-sheet/induced-abortion-worldwide

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 40cc Buffered 0.5% Lidocaine With 2 Units of Vasopressin Paracervical Block | 20cc 1% Lidocaine With 2 Units of Vasopressin Paracervical Block
Started | 57 | 57
Completed | 57 | 57
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 40cc Buffered 0.5% Lidocaine With 2 Units of Vasopressin Paracervical Block | 20cc 1% Lidocaine With 2 Units of Vasopressin Paracervical Block | Total
Number analyzed (Participants) | 57 | 57 | 114
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 57 | 114
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.1) | 31.5 (6.6) | 31.7 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 57 | 114
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 28 | 32 | 60
  Black or African American | 2 | 3 | 5
  Hispanic or Latina | 13 | 12 | 25
  Asian | 8 | 9 | 17
  Native Hawaiian or other Pacific Islander | 2 | 0 | 2
  Other or Multiracial | 4 | 1 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57 | 57 | 114
Induced Abortion vs Early Pregnancy Loss [Count of Participants; unit: Participants]
  D&C for Early Pregnancy Loss | 29 | 29 | 58
  D&C for Induced Abortion | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Pain With Cervical Dilation
Description: Distance (mm) from the left of the 100-mm Visual Analog Scale (VAS) (reflecting magnitude of pain) recorded at time of cervical dilation. Pain will be assessed using a 100 mm visual analogue scale with the anchors 0 = none, 100 mm = worst imaginable.
Time Frame: Once during the procedure on the day of recruitment, approximately one minute. During procedure at time of cervical dilation.
Population: Data missing for one participant in the 20cc group because cervical dilation was not performed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 20cc 1% Lidocaine With 2 Units of Vasopressin Paracervical Block | 40cc Buffered 0.5% Lidocaine With 2 Units of Vasopressin Paracervical Block
Number analyzed (Participants) | 56 | 57
units on a scale | 52 [35 to 62] | 45 [29 to 64]

2. Secondary Outcome: Pain With Uterine Aspiration
Description: Distance (mm) from the left of the 100-mm Visual Analog Scale (VAS) (reflecting magnitude of pain) recorded immediately after uterine aspiration. Pain will be assessed using a 100 mm visual analogue scale with the anchors 0 = none, 100 mm = worst imaginable.
Time Frame: Once during the procedure on the day of recruitment, approximately 1 minute. During procedure immediately after uterine aspiration.
Population: Data missing for one participant in the 20cc group because aspiration unable to be performed.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 20cc 1% Lidocaine With 2 Units of Vasopressin Paracervical Block | 40cc Buffered 0.5% Lidocaine With 2 Units of Vasopressin Paracervical Block
Number analyzed (Participants) | 56 | 57
units on a scale | 46 [23 to 65] | 58 [41 to 72]

3. Secondary Outcome: Pain 10 Minutes Post Procedure
Description: Distance (mm) from the left of the 100-mm Visual Analog Scale (VAS) (reflecting magnitude of pain) recorded 10 minutes after the completion of the procedure. Pain will be assessed using a 100 mm visual analogue scale with the anchors 0 = none, 100 mm = worst imaginable.
Time Frame: Once 10 minutes after the procedure on the day of recruitment, approximately one minute.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 20cc 1% Lidocaine With 2 Units of Vasopressin Paracervical Block | 40cc Buffered 0.5% Lidocaine With 2 Units of Vasopressin Paracervical Block
Number analyzed (Participants) | 57 | 57
units on a scale | 26 [6 to 50] | 11 [3 to 48]

4. Secondary Outcome: Overall Pain
Description: Distance (mm) from the left of the 100-mm Visual Analog Scale (VAS) (reflecting magnitude of pain) recorded after the procedure reflecting the overall pain felt during the procedure. Pain will be assessed using a 100 mm visual analogue scale with the anchors 0 = none, 100 mm = worst imaginable.
Time Frame: Once 10 minutes after the procedure on the day of recruitment, approximately one minute.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | 20cc 1% Lidocaine With 2 Units of Vasopressin Paracervical Block | 40cc Buffered 0.5% Lidocaine With 2 Units of Vasopressin Paracervical Block
Number analyzed (Participants) | 57 | 57
units on a scale | 57 [50 to 65] | 56 [48 to 76]

ADVERSE EVENTS:
Time Frame: From time of consent through clinical discharge time. Approximately 90 minutes.
Description: Serious adverse events: seizure or cardiac arrest. Other non-serious events: minor side effects (transient lightheadedness, tinnitus, circumoral tingling, and a metallic taste in the mouth)
Arm/Group | 20cc 1% Lidocaine With 2 Units of Vasopressin Paracervical Block | 40cc Buffered 0.5% Lidocaine With 2 Units of Vasopressin Paracervical Block
All-Cause Mortality (participants affected / at risk) | 0/57 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/57
Other Adverse Events (participants affected / at risk) | 15/57 | 12/57
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20cc 1% Lidocaine With 2 Units of Vasopressin Paracervical Block (N=57) | 40cc Buffered 0.5% Lidocaine With 2 Units of Vasopressin Paracervical Block (N=57)
Minor adverse events (Nervous system disorders) | 15 (15) | 12 (12) — Mild reactions included transient lightheadedness (dizziness), nausea, tinnitus, peri oral numbness or tingling, and metallic taste in mouth. These side effects were not analyzed individually.

LIMITATIONS AND CAVEATS:
Limitations of our study include a lack of variation in the clinical setting for which the dilation and aspiration procedures were performed (outpatient clinics at large academic centers) limiting the generalizability of the study to community care settings. The study was powered to evaluate only a 20-mm difference in pain control within each stratum of the cohort. Larger sample sizes in each stratum could potentially detect a more subtle effect on pain control.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/51/NCT03636451/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT03636451/ICF_001.pdf